CLINICAL TRIAL: NCT01551511
Title: Δ9-THC (Namisol®) in Chronic Pancreatitis Patients Suffering From Persistent Abdominal Pain: a Randomized, Double-blinded, Placebo-controlled, Parallel Design
Brief Title: Δ9-THC (Namisol®) in Chronic Pancreatitis Patients Suffering From Persistent Abdominal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HEEL-2011-02
Record Dates: First submitted 2012-02-07; First posted 2012-03-12 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Pancreatitis, Chronic; Abdominal Pain; Chronic Pain
Keywords: chronic pancreatitis; abdominal pain; visceral pain; chronic pain
MeSH Terms: conditions — Pancreatitis, Chronic; Abdominal Pain; Chronic Pain; Visceral Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- delta-9-tetrahydrocannabinol (namisol) (Experimental)
  Interventions: Drug: Tetrahydrocannabinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — The add-on treatment consists of two phases: a step-up phase (day 1-5: 3 mg TID; day 6-10: 5 mg TID), and a stable dose phase (day 11-52: 8 mg TID). The dosage may be tapered to at least 5 mg TID, when 8 mg is not tolerated.
  Other Names: Namisol; Dronabinol
  Arms: delta-9-tetrahydrocannabinol (namisol)
Drug: Placebo — Identical step-up approach to the Namisol arm.
  Arms: Placebo

SUMMARY:
Abdominal pain resulting from chronic pancreatitis (CP) is often recurrent, intense and long-lasting, and is extremely difficult to treat. Medical analgesic therapy is considered as first choice in pain management of CP, resulting in regularly prescription of opioids. The adverse consequences of prolonged opioid use, including addiction, tolerance and opioid induced hyperalgesia, call for an alternative medical treatment. Cannabis has been used to treat pain for many centuries. Delta-9-tetrahydrocannabinol (Δ9-THC), the psychoactive substance of the cannabis plant, has been shown in previous studies to be a promising analgesic. The development of Namisol®, a tablet containing purified Δ9-THC showing an improved pharmacokinetic profile, provides the opportunity to test the analgesic potential of Δ9-THC in favourable conditions. The current study aims to investigate the analgesic efficacy of Namisol® as add-on analgesic during a long-term treatment (52 days) of abdominal pain resulting from CP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed chronic pancreatitis
* Pain duration exceeding 3 months, and average NRS≥3
* Stable doses intake of analgesics for the past 2 months
* The patient has been informed about the study, understood the information and signed the informed consent form

Exclusion Criteria:

* Patient took cannabinoids on a regular basis for at least one year
* Patient does not feel a pinprick test in the lower extremities
* Patient has a body mass index (BMI) above 32,0 kg/m2
* Patient suffers from serious painful conditions other than chronic pancreatitis
* Patient has a significant medical disorder that may interfere with the study or may pose a risk for the patient
* Patient uses any kind of concomitant medication that may interfere with the study or may pose a risk for the patient
* Patient does not tolerate oral intake of medication or liquids, or is refrained from oral intake because of medical reasons
* Patient demonstrates clinical relevant deviations in the electrocardiogram (ECG)
* Patient has an actual moderate to severe renal impairment
* Patient has an actual moderate to severe hepatic impairment
* Patient has a presence or history of major psychiatric illness
* Patient has experienced an epileptic seizure in the past
* Patient demonstrates clinically significant laboratory abnormalities
* Patient demonstrates a positive urine drug screen for THC, cocaine, MDMA, and amphetamines
* Patient demonstrates a positive test result on hepatitis B surface antigen, hepatitis C antibody or HIV antibody test
* Patient has a history of sensitivity / idiosyncrasy to THC
* Patient has a known or suspected lactose intolerance
* Female patient is pregnant or breastfeeding
* Patient intends to conceive a child during the course of the study
* Patient participates in another investigational drug study
* Patient has a clinical significant exacerbation in illness
* Patient is unwilling or unable to comply with the lifestyle guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Average VAS pain | Baseline versus day 52
  The primary outcome measure is defined as the reduction in average VAS pain scores at the end of the study (day 50-52) compared to the pre-treatment level between the Namisol® and placebo group, measured by a Visual Analoge Scale (VAS) in a daily pain diary.

SECONDARY OUTCOMES:
EEG | Baseline and day 52
  Electroencephalogram; measuring evoked potentials to noxious electrical stimuli, evoked potentials to auditory stimuli (oddball), and FFT of spontaneous EEG.
QST | Baseline versus day 15 and day 52
  Quantitative Sensory Testing; measuring pressure pain thresholds, electrical thresholds, electric wind-up response, and DNIC.
Safety | Baseline until follow-up (day 59-61)
  * Laboratory
  * ECG
  * HF / BP
  * Adverse events
Pharmacokinetics | Predose levels at baseline, day 15 and day 52; postdose levels (30 min, 45 min, 60 min, 100 min) at day 15 and 52
  THC, 11-OH-THC and THC-COOH concentrations
Functional parameters | Baseline until day 52
  * Body weight
  * Supplementary feeding
Quality of life | Baseline versus day 52
  Quality of life will be evaluated by questionnaires
Pharmacodynamics | Baseline versus day 15 and day 52
  Pharmacodynamics measured by body sway and questionnaires (VASBond & Lader and VASBowdle)

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, department of surgery
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] de Vries M, van Rijckevorsel DCM, Vissers KCP, Wilder-Smith OHG, van Goor H; Pain and Nociception Neuroscience Research Group. Tetrahydrocannabinol Does Not Reduce Pain in Patients With Chronic Abdominal Pain in a Phase 2 Placebo-controlled Study. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1079-1086.e4. doi: 10.1016/j.cgh.2016.09.147. Epub 2016 Oct 5. PMID 27720917